CLINICAL TRIAL: NCT05109208
Title: Ultrasound Vibroelastography in Post-Prostatectomy Erectile Dysfunction
Brief Title: The Use of Ultrasound in Assessing Post-prostatectomy Erectile Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew (Matt) J. Ziegelmann, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-001713; NCI-2024-00502 (Other Grant/Funding Number: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Prostate Adenocarcinoma
Keywords: Radical Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrasound viscoelastography (UVE) in radical proctectomy recovery (Experimental): Subjects undergoing radical prostatectomy for prostate cancer disease as standard of care will have a ultrasound vibroelastography performed before surgery, 3 months, 6 months and 9 months post-prostatectomy.
  Interventions: Diagnostic Test: Ulrasound Vibroelastography (UVE)

INTERVENTIONS:
Diagnostic Test: Ulrasound Vibroelastography (UVE) — Ultrasound technique to quantitatively assess tissue stiffness (elasticity and viscosity) by applying vibration through a specialized probe (indenter).

SUMMARY:
Researchers are trying to determine whether there is additional utility to using vibroelastography, a noninvasive ultrasound technique to evaluate for the presence of tissue fibrosis, in conjunction with standard penile duplex Doppler ultrasound to assess erectile function (recovery) after prostate cancer surgery.

ELIGIBILITY:
Inclusion criteria include:

* Age > 40 years
* Clinically localized prostate cancer (American Urological Association Grade Groups 1-2; cT1c or cT2a-b; PSA < 10) without clinic or imaging evidence of localized extra-prostatic or metastatic disease (i.e. AUA low and favorable intermediate risk prostate cancer)
* International Index of Erectile Function (IIEF) of ≥ 21 points at baseline (no or mild erectile dysfunction)
* Patient-expressed interest in consultation for sexual function (erectile function) preservation/ optimization
* Planned bilateral nerves-paring prostatectomy

Exclusion criteria include:

* Moderate or severe ED based in IIEF criteria (score < 21)
* History of prior pelvic or penile surgery
* Current or prior androgen deprivation therapy
* Planned non-nerve sparing prostatectomy

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in Viscoelasticity | Baseline, 3 months, 6 months and 9 months post-prostatectomy
  As measured by Ultrasound Vibroelastography (UVE)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Ziegelmann, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials